CLINICAL TRIAL: NCT05511701
Title: Preventing Ischemic Heart Disease With mHealth, Electronic Decision Support, and Community Health Workers (PRIMECare Trial)
Brief Title: Preventing Ischemic Heart Disease With mHealth (Mobile Health), Electronic Decision Support and Community Health Workers
Acronym: PRIMECare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Thomas Gaziano, Associate Professor, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-1166
Record Dates: First submitted 2022-08-05; First posted 2022-08-23 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases (CVD)
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): with paper-based guidelines used by community health workers (CHW) and providers
  Interventions: Behavioral: Usual Care Model
- Intervention (Experimental): with central data management system linking digital mHealth screening tool for CHWs, electronic appointment scheduling, point of care testing (POCT) for lipids, clinical decision support for medication initiation, and a SMS reminder system for adherence to medications and life-style changes
  Interventions: Behavioral: CHW Care Model

INTERVENTIONS:
Behavioral: CHW Care Model — The CHW will measure the participant's blood pressure (BP) and along with other demographic variables, calculate the participant's absolute CVD risk score, using the mHealth (mobile health) app. If the participant's risk is > 10%, they are asked to sign the informed consent. The CHW will electronically schedule an appointment at the PCC. The participant will receive a SMS appointment confirmation. S/he will have their cholesterol tested by nurses using a home POCT. Nurses will repeat POCT lipids and BP measurements at all PCC visits and other clinical information will be entered into the electronic decision support tool that will generate a guideline based treatment recommendation for the physician. CHWs will make up to four home visits or telephone calls to intervention participants over the 12 month study period to check on medication adherence, as well as to determine if the patient is in possession of the medication
  Arms: Intervention
Behavioral: Usual Care Model — All study participants will be visited in their home by a CHW and a nurse for eligibility assessment, screening, and enrollment. The CHW will then measure the participant's blood pressure and the readings along with other demographic variables already collected, to calculate the participant's absolute CVD risk score. In the usual care arm the CHW will use the WHO paper-based non-lab CVD risk calculator and, if the participant's risk is > 10%, they are asked to sign the informed consent and s/he will have their cholesterol tested by nurses using POCT during a home enrollment visit. The CHW will further verbally encourage her/him to schedule an appointment with a primary care physician at the PCC for evaluation. This is the usual care practice.
  Arms: Usual Care

SUMMARY:
This is a cluster-randomized clinical trial (cRCT) designed to assess the effectiveness of a multicomponent strategy linking key aspects of the cardiovascular disease (CVD) care continuum across three provinces in Argentina using using five primary components: a data management system linking a digital mHealth (mobile health) screening tool used by community health workers (CHWs), an electronic appointment scheduler which is integrated with the clinic electronic appointment system, point of care (POCT) testing for lipids, a clinical decision support system for medication initiation, and a text message (SMS) reminder system to improve treatment adherence and life-style changes.

DETAILED DESCRIPTION:
954 eligible women and men aged 40-74 with high CVD risk living in the catchment area of 18 primary care clinics (PCCs) in 3 different provinces (Quilmes, La Rioja, and San Juan) in Argentina will be recruited for the study. Eighteen PCCs will be randomized to either the usual care (control) arm or the intervention arm (3 usual care and 3 intervention PCCs in each province). Participants who reside in the catchment area of intervention PCCs will receive the multicomponent intervention with central data management system linking digital mHealth (mobile health) screening tool for CHWs, electronic appointment scheduling which is integrated with the clinic electronic appointment system, point of care testing (POCT) for lipids, clinical decision support for medication initiation, and a SMS reminder system for adherence to medications and life-style changes, while participants who reside in the catchment area of usual care PCCs will receive usual care with paper-based guidelines used by community health workers and providers. The recruitment goals are 477 persons in the intervention arm and 477 in the usual care arm. Participants will be enrolled for a 12 month study period from baseline visit, and the primary outcome is mean difference in absolute 10-year CVD risk.

ELIGIBILITY:
Inclusion Criteria:

* aged 40-74
* depend exclusively on public health insurance
* have access to a cell phone for personal use
* can open and read SMS messages on cell phone
* receive primary care at the local PCC
* have a 10-year CVD risk >= 10% and mean SBP >= 140 mmHg OR
* have a 10-year CVD risk >= 10% and LDL-C >= 70 mg/dL for persons with diabetes OR
* have a 10-year CVD risk >= 10% and LDL-C >= 100 mg/dL for persons without diabetes

Exclusion Criteria:

* Persons who plan to move from the neighborhood within the next 2 years
* pregnant at the time of screening
* Bed bound
* Weight > 180 kg - this exceeds the upper limit that can be measured on portable scales.
* Total cholesterol < 100 mg/dL or > 500 mg/dL.
* LDL-C > 300 mg/dL
* Triglycerides < 45 mg/dL or > 400 mg/dL.
* HDL < 15 mg/dL.
* Systolic blood pressure (SBP) >=180 mmHg or Diastolic blood pressure (DBP) >= 120 mmHg, and experiencing chest pain, palpitations, or shortness of breath.
* currently on dialysis or has a history of chronic kidney disease.
* self-reported history of CVD (stroke, AMI).
* self-reported history of a liver abnormality.
* have a mid-upper arm circumference > 42 cm - this is the maximum cuff size available for use with blood pressure monitors in Argentina
* do not consent to participate.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 954 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Difference in mean change in absolute CVD risk, calculated using the Framingham cardiovascular disease lab-based risk equation, between study arms at 12 months | At enrollment (baseline) and 12 months after enrollment
  The difference in mean change in 10-year CVD risk between study arms

SECONDARY OUTCOMES:
Difference in mean change in LDL-C between study arms at 12 months | At enrollment (baseline) and 12 months after enrollment
  The difference in mean change in LDL-C between study arms.
Difference in mean change in systolic blood pressure between study arms at 12 months | At enrollment (baseline) and 12 months after enrollment
  The difference in mean change in systolic blood pressure between study arms.
Changes in smoking rates over 12-month study period | At enrollment (baseline) and 12 months after enrollment
  The difference in mean smoking rates between study arms
Medical costs incurred over 12-month study period | From enrollment to end of the study period at 12 months
  The difference in medical costs between study arms
Medication possession ratios at 12 months between study arms | At 12 months after enrollment
  Ratio of prescribed statins and anti-hypertension medications in participants' possession
Medication intensity changes | From enrollment to end of the study period at 12 months
  Number of treatment intensity changes for statins and anti-hypertension medications in the intervention arm
Major adverse reactions for statins and anti-hypertension medications | From enrollment to end of the study period at 12 months
  Number of reported adverse reactions for statins and anti-hypertension medications in intervention arm
Quality adjusted life years (QALYs) | From enrollment to end of the study period at 12 months
  Summary of the impact the intervention on CVD risk
Proportion of patients with a 10-year CVD risk ≥ 10% that complete a first visit at the local clinic within 6 weeks after enrollment in the study. | 6 weeks from enrollment.
  Proportion of patients with a 10-year CVD risk ≥ 10% that complete a visit at the local clinic within 6 weeks after enrollment in the study.
Proportion of patients with a 10-year CVD risk ≥ 10% that complete a first visit at the local clinic within 4 months after enrollment in the study. | 4 months from enrollment
  Proportion of patients with a 10-year CVD risk ≥ 10% that complete a first visit at the local clinic within 4 months after enrollment in the study.
Number of clinical visits between study arms at 12 months | From enrollment to end of the study period at 12 months
  Number of clinical visits by participants to primary care clinics
Health utilization outcomes | From enrollment to end of the study period at 12 months
  Number of hospitalizations, emergency room visits, outpatient visits and procedures, and primary care clinic visits
Mortality | From the start of enrollment to 12, then 60 months after enrollment
  Number of deaths from all causes

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Gaziano, MD, MSc, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Iecs Instituto de Efectividad Clinica Y Sanitaria, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Because of the sensitive nature of the data collected for this study, requests to access the data set from qualified researchers trained in human subject confidentiality protocols may be sent to the primary investigator.
Supporting Information: Study Protocol, ICF
Time Frame: After the date of study closure up to 5 years.
Access Criteria: Investigators who wish to use the data will be required to send a detailed proposal, including an analytic plan, to the primary investigator for review.

DOCUMENTS (1):
  • Informed Consent Form (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT05511701/ICF_000.pdf